CLINICAL TRIAL: NCT04143763
Title: The Effect of an Ecological Momentary Intervention for Stroke Caregivers' Psychological Support: a Pilot Feasibility Trial
Brief Title: Mobile Message Intervention for Stroke Caregivers' Psychological Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jung-Jae Lee, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HKUSON_LEE1
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Stroke; Caregiver Burnout; Mobile Phone Use; Depressive Symptoms; Psychological Distress
MeSH Terms: conditions — Stroke; Caregiver Burden; Cell Phone Use; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): receive mobile messages supporting caregivers' psychological well-being, according to the participants' preferences in intervention group.
  Interventions: Other: Ecological Momentary Intervention (EMI)
- Control group (No Intervention): receive general health information through a mobile message.

INTERVENTIONS:
Other: Ecological Momentary Intervention (EMI) — Using the messaging function of mobile devices, EMI offers a framework to deliver health information to the target population, corresponding to each individual's demands in terms of type (e.g., photo, text and/or voice message), timing, duration, and frequency of the messages, which are different to the features from other interventions
  Arms: Intervention group

SUMMARY:
The proposed trial aims to test the feasibility of ecological momentary intervention on stroke caregivers' psychological distress.

DETAILED DESCRIPTION:
75% of stroke caregivers report severe caregiver burdens, with 60% of stroke caregivers reporting at least one depressive symptom in Hong Kong. However, caregivers can experience difficulties in accessing and fully utilising existing services due to the varying types of care needs and its intensities amongst stroke survivors.

Ecological momentary intervention (EMI) as an innovative and personalised intervention has shown great potential in supporting psychological well-being; yet, there are no studies on using EMI for the caregivers' psychological support. The proposed trial aims to reduce stroke caregivers' psychological distress by delivering EMI through instant messaging applications to provide personalised and real-time support led by healthcare professionals.

Stroke caregivers screened by Patient Health Questionnaire-9 (PHQ-9) with scores ranging from 5 to 19 will be recruited from multiple sites including community centres, rehabilitation centres and outpatient clinics in public hospitals in Hong Kong, and individually randomised into the intervention group (n=20) or control group (n=20). The intervention group will receive the personalised instant messages for 4 weeks. The control group will receive general health information and regular messages reminding them to participate in follow-up surveys. The primary outcome will be the score of PHQ-9 at 4 weeks. Secondary outcomes will include anxiety, perceived stress, and caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* Primary family caregiver of stroke survivor
* Able to read and communicate in Chinese
* Able to use mobile phone text messaging function
* PHQ-9 ranged from 5 to 19

Exclusion Criteria:

* Professional medical personnel and care assistants
* Has provided care for <1 month prior to recruitment
* Has diagnosis of psychiatric disease or is currently taking psychotropic drug
* PHQ-9 ≥ 20 (i.e., severe depressive symptom)
* Currently participating in any type of psychological support intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Change depressive symptoms by Patient Health Questionnaire (PHQ-9) Scale (questionnaire) at 4 weeks | 4 weeks
  Patient Health Questionnaire (PHQ-9) Scale: PHQ-9 is a scale for screening depression in primary care. It consists of 9 items with 4 likert scale. Score range is from 0 to 27 (higher score = higher severity of depressive symptom).

SECONDARY OUTCOMES:
Change anxiety symptoms by Generalized Anxiety Disorder-7 (GAD-7) Scale at 4 weeks | 4 weeks
  Generalized Anxiety Disorder-7 (GAD-7) Scale: GAD-7 is a scale for screening anxiety in primary care. It consists of 7 items with 4 likert scale.
  Score range is from 0 to 21 (higher score = higher severity of anxiety symptom).
Change stress levels by Perceived Stress Scale (PSS-4) at 4 weeks | 4 weeks
  Perceived Stress Scale (PSS-4); PSS-4 is a scale for screening stress level. It consists of 4 items with 5 likert scale. Score range is from 0 to 16 (higher score = higher severity of stress).
Change caring burdens by Burden Interview-4 (ZBI-4) at 4 weeks | 4 weeks
  Burden Interview-4 (ZBI-4) Scale: ZBI-4 is a scale for screening carer's burdens. It consists of 4 items with 5 likert scale.
  Score range is from 0 to 16 (higher score = higher severity of caring burden).

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Hong Kong PHAB Association, Hong Kong
  - Hong Kong Stroke Association, Hong Kong

IPD SHARING:
Plan to Share IPD: No